CLINICAL TRIAL: NCT03557320
Title: Impact of Meteorological Conditions on the Onset of First Episod of Spontaneous Pneumothorax : a French Multicenter Case-crosserover Study About 945 Subjects in 14 Centers
Brief Title: Environmental Factor and Onset of Spontaneous Pneumothorax
Acronym: EXPPO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); Centre Hospitalier Universitaire Dijon (Other); Hopital Nord Franche-Comte (Other); Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other); Centre Hospitalier de la Haute Saone (Unknown); CHU de Reims (Other); Centre Hospitalier de Bethune (Network); Centre Hospitalier Saint Philibert Lomme (Unknown); Centre Hospitalier de Roubaix (Other); Boulogne sur Mer Hospital Center (Other); Poitiers University Hospital (Other); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Universitaire de Angers (Unknown); Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: API/2012/29
Record Dates: First submitted 2016-09-05; First posted 2018-06-15 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Spontaneous Pneumothorax
Keywords: environment; pressure; temperature; case-crossover
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the association between spontaneous pneumothorax onset and weather parameters.

DETAILED DESCRIPTION:
The aim of this study is to analyse the relation between onset of the PSP and exposure to environmental factors such as atmospheric pressure.

A case-crossover epidemiological study will be conducted in 14 French hospitals. SP recorded from 2009 to 2013 will be exhaustively included. Demographic and clinical characteristics will be collected. For each incident case of SP, the period of occurrence of the event (case period) will be compared to several other periods temporally distant from the case period (control periods prior to and after the event). Exposure will be assessed using meteorological stations localized in the vicinity of each patient's home. A potential threshold effect and/or time lag effect between exposure and admission for SP will be explored.

The results of this study will help to identify the meteorological factors associated with the occurrence of SP, and to deepen our knowledge of the pathophysiological mechanisms of SP especially the influence of meteorological factors on bleb rupture.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* first episode of primary spontaneous pneumothorax

Exclusion Criteria:

* Patients with traumatic
* Patients with secondary pneumothorax
* Patients with recurrent pneumothorax and patients with short-term readmissions (recurrence was defined as a new ED admission for the same diagnosis more than 14 days after the first admission).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited in the emergency departments (ED) of fourteen French hospitals that are members of the EXPRED Network (EXPRED Study) (Desmettre et al. 2011) where emergency admission management software was available.
  A search was performed of ED admissions databases to identify all patients with a primary diagnosis of pneumothorax (International Classification of Diseases (ICD) 10 code = J93) admitted between June 1, 2009 and May 31, 2013).
Sampling Method: Non-Probability Sample
Enrollment: 3090 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Estimate odds ratio for the association between meteorological data and onset of PSP. | 28 days

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Angers, Angers
  - Centre Hospitalier de Belfort, Belfort
  - CH Boulogne sur Mer, Boulogne-sur-Mer
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - Polyclinique de DIVION, Divion
  - Clinique de HENIN BEAUMONT, Hénin-Beaumont
  - CH Lomme, Lomme
  - CH Mulhouse, Mulhouse
  - CHU Nimes, Nîmes
  - CHU Poitiers, Poitiers
  - CHU Toulouse, Toulouse
  - Centre Hospitalier de Vesoul, Vesoul

IPD SHARING:
Plan to Share IPD: No